CLINICAL TRIAL: NCT00485134
Title: Shigella Flexneri 2a Invaplex 50 Vaccine Dose Finding and Assessment of Protection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: U.S. Army Office of the Surgeon General (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NMRC.2006.0007; HSRRB # A-14057 (Other: USAMRMC); WRAIR 1328 (Other: Walter Reed Army Institute of Research)
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Stage 1: Group A, Dolphin 240 µg (Experimental): 240 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of lipopolysaccharides (LPS). 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (DolphinTM).
  Interventions: Biological: 240 µg Shigella flexneri 2a Invaplex 50 vaccine
- Stage 1: Group B, Dolphin 480 µg (Experimental): 480 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (DolphinTM).
  Interventions: Biological: 480 µg Shigella flexneri 2a Invaplex 50 vaccine
- Stage 1: Group C, Dolphin 690 µg (Experimental): 690 Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (DolphinTM).
  Interventions: Biological: 690 Shigella flexneri 2a Invaplex 50 vaccine
- Stage 1: Group D, Pipette 240 µg (Other): 240 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. These subjects received 200 μL the vaccine via electronic pipette. This group is for lot bridging only, not included in dose-finding study.
  Interventions: Biological: 240 µg Shigella flexneri 2a Invaplex 50 vaccine
- Stage 2: Immunized / Challenge (Other): The selected dose was to be administered with the Dolphin™ using the vaccination schedule from stage 1. Immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Interventions: Other: Shigella challenge strain
- Stage 2: Controls (Placebo Comparator): A control was to be administered with the DolphinTM using the vaccination schedule from Stage 1. Non-immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Interventions: Other: Shigella challenge strain

INTERVENTIONS:
Biological: 240 µg Shigella flexneri 2a Invaplex 50 vaccine — Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
  Arms: Stage 1: Group A, Dolphin 240 µg; Stage 1: Group D, Pipette 240 µg
Biological: 480 µg Shigella flexneri 2a Invaplex 50 vaccine — Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
  Arms: Stage 1: Group B, Dolphin 480 µg
Biological: 690 Shigella flexneri 2a Invaplex 50 vaccine — Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
  Arms: Stage 1: Group C, Dolphin 690 µg
Other: Shigella challenge strain — 300 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T
  Other Names: Shigella challenge material
  Arms: Stage 2: Controls; Stage 2: Immunized / Challenge

SUMMARY:
The purpose of this study is to select a safe and immunogenic dose of Invaplex 50 intranasal vaccine, and to assess protection of Invaplex 50 intranasal vaccine against diarrhea, dysentery, and fever following challenge with the Shigella flexneri 2a 2457T strain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved ≥ 70% accuracy).
* Signed informed consent form.
* Available for the required follow-up period and scheduled clinic visits.
* Women: negative pregnancy test with understanding (through informed consent process) to not become pregnant during the study or within two (2) months following study completion.

Exclusion Criteria:

General Health

* Health problems affecting study participation from medical history specifically to include chronic medical conditions such as psychiatric conditions, diabetes mellitus and hypertension or any other condition requiring chronic daily therapy that would place the volunteer at increased risk - as determined by a study physician, current use of antihypertensive medications, or other medications that may interact with pseudoephedrine in the event it is required to treat rhinorrhea).
* Clinically significant abnormalities on physical examination.
* Use of immunosuppressive drugs such as corticosteroids or chemotherapeutics that may influence antibody development.
* Women currently nursing
* Participation in research involving another investigational product (defined as receipt of investigational product or exposure to invasive investigational device) 30 days before planned date of first vaccination or anytime throughout the duration of the study.
* Positive blood test for HBsAG, HCV, HIV-1.
* Clinically significant abnormalities on basic laboratory screening.
* Immunosuppressive illness or IgA deficiency (below the normal limits).

Research specific

* Presence of nasal polyps, ulcers, or deviated nasal septum (further defined in section 4.2).
* History of chronic sinusitis or chronic/seasonal rhinitis (further defined in section 4.2)
* History of rhinoplasty.
* History of reactive airway disease (asthma), chronic obstructive pulmonary disease, or chronic bronchitis.
* History of Bell's palsy.
* Current smoker or smoker in past 3 months ('smoker' defined as daily cigarette cigar, or pipe use for a period of at least 1 month).
* Regular use (weekly or more often of antidiarrheal, anti-constipation, or antacid therapy
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
* Personal or family history of an inflammatory arthritis.
* Positive blood test for HLA-B27.
* Prior exposure to Shigella
* History of microbiologically confirmed Shigella infection.
* Received previous experimental Shigella vaccine or live Shigella challenge.
* Travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within two years prior to dosing.
* Occupation involving handling of Shigella bacteria currently, or in the past 3 years.
* Serum IgG titer ≥ 2500 to Shigella LPS

Additionally, subjects participating in stage 2 with any of the following will be excluded:

* Are employed as a food handler, daycare provider or work in a nursing home, or are in direct care of an immunocompromised person, a child <2 years of age or frail elderly.
* Significant abnormalities in pre-admission screening lab hematology, serum chemistry, urinalysis or EKG (EKG only in volunteers ≥40 years), as determined by PI or the PI in consultation with the medical monitor and sponsor.
* Allergy to ciprofloxacin on ampicillin (excluded if allergic to either).
* History of diarrhea in the 2 weeks prior to planned inpatient phase.
* Use of antibiotics during the 7 days before Shigella inoculation or proton pump inhibitors, H2 blockers, or antacids within 48 hours of inoculation.
* Inability to comply with inpatient rules and regulations.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Riddle, MD, Principal Investigator — Naval Medical Research Center
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR) John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Department of Clinical Trials, WRAIR, Silver Spring, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: Group A, Dolphin 240 µg: 240 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of lipopolysaccharides (LPS). 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (Dolphin™).
  240 µg Shigella flexneri 2a Invaplex 50 vaccine: Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
- Stage 1: Group B, Dolphin 480 µg: 480 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (Dolphin™).
  480 µg Shigella flexneri 2a Invaplex 50 vaccine: Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
- Stage 1: Group C, Dolphin 690 µg: 690 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (Dolphin™).
  690 µg Shigella flexneri 2a Invaplex 50 vaccine: Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
- Stage 2: Dolphin 690 ug (CTC WRAIR Site); Stage 2: Dolphin 690 ug (JHU CIR Site): 690 ug shigella flexneri 2a Invaplex 50 was to be administered with the Dolphin™ using the vaccination schedule from stage 1. Immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Some individuals were randomly selected for the challenge phase. Shigella challenge strain: 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T
- Stage 2: Placebo Group (CTC WRAIR Site): Stage 2: Placebo group (CTC WRAIR site) A control was to be administered with the Dolphin™ using the vaccination schedule from Stage 1. Non-immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Some individuals were randomly selected for the challenge phase. Shigella challenge strain: 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T
- Stage 2: Placebo Group (JHU CIR Site): A control was to be administered with the Dolphin™ using the vaccination schedule from Stage 1. Non-immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Some individuals were randomly selected for the challenge phase. Shigella challenge strain: 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T
Period: Overall Study
Arm/Group | Stage 1: Group A, Dolphin 240 µg | Stage 1: Group B, Dolphin 480 µg | Stage 1: Group C, Dolphin 690 µg | Stage 1: Group D, Pipette 240 µg | Stage 2: Dolphin 690 ug (CTC WRAIR Site) | Stage 2: Placebo Group (CTC WRAIR Site) | Stage 2: Dolphin 690 ug (JHU CIR Site) | Stage 2: Placebo Group (JHU CIR Site)
Started | 12 | 12 | 12 | 8 | 10 | 7 | 31 | 21
Completed | 11 | 10 | 9 | 7 | 7 | 3 | 28 | 20
Not Completed | 1 | 2 | 3 | 1 | 3 | 4 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Change in health status | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrew for adverse event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Positive drug test | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Not completed — Unable to comply with study schedule | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stage 1: Group A, Dolphin 240 µg: 240 µg Shigella flexneri 2a Invaplex 50 vaccine. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 mL glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. 230 μL of the formulated vaccine (or placebo, sterile saline) was added to a nasal spray applicator (Dolphin™).
  240 µg Shigella flexneri 2a Invaplex 50 vaccine: Vaccines were administered intranasally on Days 0, 14, and 28. The investigational vaccine was supplied as 1 mL of a sterile, clear liquid in a 3 ml glass vial. Each vial contained 3.5 mg of protein and 567 μg of LPS. The pH was 8.9 and the buffer was 250 mM NaCl in 20 mM Tris.
- Stage 2: Placebo Group (CTC WRAIR Site); Stage 2: Placebo Group (JHU CIR Site): A control was to be administered with the Dolphin™ using the vaccination schedule from Stage 1. Non-immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Some individuals were randomly selected for the challenge phase. Shigella challenge strain: 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T
- Total: Total of all reporting groups
Arm/Group | Stage 1: Group A, Dolphin 240 µg | Stage 1: Group B, Dolphin 480 µg | Stage 1: Group C, Dolphin 690 µg | Stage 1: Group D, Pipette 240 µg | Stage 2: Dolphin 690 ug (CTC WRAIR Site) | Stage 2: Placebo Group (CTC WRAIR Site) | Stage 2: Dolphin 690 ug (JHU CIR Site) | Stage 2: Placebo Group (JHU CIR Site) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 8 | 10 | 7 | 31 | 21 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] — Age for stage 2 groups do not include data from individuals who were at Walter Reed Army Institute of Research (WRAIR) Clinical Trials Center (CTC) (10 immunized and 7 controls). Data is entered as presented in the Final Clinical Study Report.
  years | 38.1 (7.1) | 39.6 (4.4) | 30.7 (7.3) | 29.3 (7.1) | 35.1 (10.2) | 34.4 (10.4) | 32.2 (8.3) | 31.3 (8.2) | 33.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 3 | 4 | 2 | 13 | 15 | 54
  Male | 7 | 7 | 5 | 5 | 6 | 5 | 18 | 6 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 7 | 8 | 9 | 2 | 6 | 6 | 27 | 17 | 82
  Caucasian | 5 | 3 | 1 | 3 | 1 | 1 | 3 | 4 | 21
  Other | 0 | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 8
  Data Missing | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Post-challenge Diarrhea, Fever, and Blood in Stool Adverse Events by Study Group
Description: Fecal samples were collected through day 77 or until discharge (all stools collected for weighing/grading; maximum of 3 stools/day for culture; rectal swab obtained if no stool provided).
Time Frame: 7 days after challenge
Population: The decision criteria to progress to challenge with the Shigella challenge strain were no limiting adverse events (AEs) and positive immune response. These individuals were challenged with 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T.
Measure: Number; unit: participants
Groups:
- Stage 2: Controls: A control was to be administered with the Dolphin™ using the vaccination schedule from Stage 1. Non-immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Some individuals were randomly selected for the challenge phase. Shigella challenge strain: 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T.
- Stage 2: Immunized: The selected dose was to be administered with the Dolphin™ using the vaccination schedule from stage 1. Immunized and challenged with Shigella challenge strain approximately 42 days after receiving the last vaccination following a 90-minute fast.
  Some individuals were randomly selected for the challenge phase. Shigella challenge strain: 800 colony forming units (CFU) of Shigella challenge strain, Shigella flexneri 2a strain 2457T.
Arm/Group | Stage 2: Controls | Stage 2: Immunized
Number analyzed (Participants) | 12 | 10
participants
  Mild diarrhea | 1 | 0
  Moderate diarrhea | 4 | 4
  Severe diarrhea | 3 | 3
  Fever | 4 | 5
  Blood in stools | 4 | 5

2. Secondary Outcome: Post-challenge Loose Stool Samples Occurrences by Study Group
Time Frame: 7 days after challenge
Population: One subject in each group had diarrhea continuing at discharge so measured stool output likely an underestimate.
Measure: Mean (Full Range); unit: loose stools
Arm/Group | Stage 2: Controls | Stage 2: Immunized
Number analyzed (Participants) | 12 | 10
loose stools
  Number of loose stools | 6.5 [4.0 to 8.0] | 8.0 [7.0 to 13.0]
  Maximum number in 24 hours period | 4.0 [4.0 to 6.0] | 5.0 [4.0 to 9.0]

3. Secondary Outcome: Post-challenge Loose Stool Sample Volumes by Study Group
Time Frame: 7 days after challenge
Population: One subject in each group had diarrhea continuing at discharge so measured stool output likely an underestimate.
Measure: Mean (Full Range); unit: mL
Arm/Group | Stage 2: Controls | Stage 2: Immunized
Number analyzed (Participants) | 12 | 10
mL
  Total volume | 540.5 [180.5 to 1251.0] | 706.0 [537.0 to 794.0]
  Maximum volume loose stools in 24 hour period | 422.0 [180.5 to 666.5] | 492.0 [410.0 to 555.0]

4. Secondary Outcome: Post-challenge Loose Stool Sample Durations by Study Group
Time Frame: 7 days after challenge
Population: One subject in each group had diarrhea continuing at discharge so measured stool output likely an underestimate.
Measure: Mean (Full Range); unit: hours
Arm/Group | Stage 2: Controls | Stage 2: Immunized
Number analyzed (Participants) | 12 | 10
hours
  Hours to first loose stool | 59.7 [52.7 to 65.4] | 75.9 [46.0 to 90.1]
  Diarrhea duration | 32.3 [18.3 to 53.0] | 47.4 [29.3 to 63.0]

5. Secondary Outcome: S. Flexneri 2a Related Non-diarrheal Clinical Outcomes by Study Group
Time Frame: 56 days post-challenge
Measure: Number; unit: participants
Arm/Group | Stage 2: Controls | Stage 2: Immunized
Number analyzed (Participants) | 12 | 10
participants
  Nausea | 4 | 4
  Vomiting | 2 | 2
  Abdominal pain/cramps | 7 | 8
  Malaise | 5 | 5
  Bloating | 3 | 6
  Flatulence | 6 | 5
  Headache | 7 | 6
  Lightheadedness | 1 | 0
  Constipation | 0 | 0
  Abdominal tenderness | 2 | 1

6. Secondary Outcome: Number of Subjects Exhibiting an Immune Response to Invaplex 50 and/or LPS
Description: Immune responder is defined as someone with both a serologic and an ASC response to either Invaplex 50 or LPS. Immune response defined as Serology: ≥ 4-fold increase in baseline serum titer antibody cecreting cells (ASC): ≥ 10 ASC per 106 peripheral blood mononuclear cells(PBMC).
Time Frame: 56 days post-vaccination in stage 1
Population: This analysis is limited to groups A-C only and subjects receiving at least 2 doses of S. flexneri 2a Invaplex 50 or LPS
Measure: Number; unit: participants
Arm/Group | Stage 1: Group A, Dolphin 240 µg | Stage 1: Group B, Dolphin 480 µg | Stage 1: Group C, Dolphin 690 µg
Number analyzed (Participants) | 11 | 10 | 12
participants | 3 | 2 | 7

ADVERSE EVENTS:
Time Frame: Subjects Participating in Stages 1 and 2 who Experienced Surveyed Signs and Symptoms Post-vaccination
Description: Group D was not included in findings due to they were for lot bridging only and not for dose-finding study.
Arm/Group | Stage 1: Group A, Dolphin 240 µg | Stage 1: Group B, Dolphin 480 µg | Stage 1: Group C, Dolphin 690 µg | Stage 2: Immunized | Stage 2: Controls
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/41 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/41 | 1/28
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12 | 11/12 | 41/41 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Group A, Dolphin 240 µg (N=12) | Stage 1: Group B, Dolphin 480 µg (N=12) | Stage 1: Group C, Dolphin 690 µg (N=12) | Stage 2: Immunized (N=41) | Stage 2: Controls (N=28)
Pregnancy (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Group A, Dolphin 240 µg (N=12) | Stage 1: Group B, Dolphin 480 µg (N=12) | Stage 1: Group C, Dolphin 690 µg (N=12) | Stage 2: Immunized (N=41) | Stage 2: Controls (N=28)
Malaise (General disorders) | 1 | 0 | 1 | 6 | 2
Headache (General disorders) | 1 | 1 | 2 | 8 | 9
Rhinorrhea (General disorders) | 4 | 3 | 4 | 10 | 9
Nasal congestion (General disorders) | 7 | 2 | 3 | 12 | 10
Nasal burning (General disorders) | 1 | 0 | 0 | 8 | 2
Nasal itching (Gastrointestinal disorders) | 1 | 4 | 5 | 5 | 0
Sore throat (General disorders) | 2 | 0 | 4 | 9 | 7
Postnasal drip (General disorders) | 2 | 2 | 5 | 8 | 6
Cough (General disorders) | 1 | 0 | 4 | 4 | 3
Sinus pain (General disorders) | 0 | 0 | 1 | 5 | 1
Sneezing (General disorders) | 1 | 4 | 5 | 14 | 4
Itching eyes (Eye disorders) | 1 | 1 | 2 | 5 | 3
Nose bleed (General disorders) | 0 | 0 | 0 | 2 | 0
Fever (General disorders) | 1 | 0 | 1 | 4 | 1
Nasal mucosa hyperemia (General disorders) | 1 | 0 | 0 | 20 | 12
Nasal discharge (General disorders) | 1 | 0 | 0 | 15 | 12
Nasal edema (General disorders) | 1 | 0 | 0 | 10 | 7
Pharyngeal erythema (General disorders) | 0 | 0 | 2 | 2 | 3
Sinus tenderness (General disorders) | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (General disorders) | 2 | 2 | 1 | 3 | 1
Conjunctival injection (Eye disorders) | 0 | 0 | 0 | 7 | 8
Tearing (General disorders) | 0 | 0 | 0 | 0 | 0
Epistaxis (General disorders) | 0 | 0 | 0 | 0 | 0
Abnormal lung exam (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Abnormal cranial nerve finding (General disorders) | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No